CLINICAL TRIAL: NCT02524587
Title: Study of the Wear of a Highly Cross-linked Polyethylene Acetabular Doped With Vitamin E and Coated With Titanium in Total Hip Replacement
Acronym: POLYTITAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-113
Record Dates: First submitted 2015-08-06; First posted 2015-08-17 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Total Hip Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- acetabular polyethylene vitamys® (Active Comparator): acetabular polyethylene vitamys®
  Interventions: Other: radio stereometric analysis (RSA) of the acetabular; Device: acetabular polyethylene vitamys®
- standard polyethylene acetabular irradiated at 3 Mrad (Active Comparator): standard polyethylene acetabular irradiated at 3 Mrad
  Interventions: Device: standard polyethylene acetabular irradiated at 3 Mrad; Other: radio stereometric analysis (RSA) of the acetabular

INTERVENTIONS:
Device: standard polyethylene acetabular irradiated at 3 Mrad
  Arms: standard polyethylene acetabular irradiated at 3 Mrad
Other: radio stereometric analysis (RSA) of the acetabular
Device: acetabular polyethylene vitamys®
  Arms: acetabular polyethylene vitamys®

SUMMARY:
The total hip replacement, with over 120,000 cases per year in France, provides short term, excellent functional results and a significant improvement in quality of life, in almost all cases. However, the observation has shown that the lifetime of the implants is limited due to aseptic loosening. One of the factors associated with these failures is a peri-prosthetic osteolysis wherein the polyethylene wear debris (PE) have been implicated. Several solutions have been proposed: change the friction torque (hard-hard pairs using ceramic or metal on the two components of the couple) or improving quality polyethylene. Improving the resistance of polyethylene wear is the primary objective evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* patients aged men and women 18 to 75 years
* with a primary or secondary osteoarthritis or osteonecrosis
* having a functional disorder requiring the installation of a total hip prosthesis of primary

Exclusion Criteria:

* patients aged 76 years or more
* pregnant or desiring to be for the duration of the study
* minors or adults protected
* repeated hip replacement
* cephalic prosthesis recovery or intermediate
* repeated cupules
* primary or secondary malignant tumor of the hip

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
penetration of the metal femoral head in acetabular | 2 years
  head penetration in milimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Département d'orthopédie - traumatologie, CHU de Caen, Caen, France

REFERENCES:
- [Derived] Rochcongar G, Remazeilles M, Bourroux E, Dunet J, Chapus V, Feron M, Praz C, Buia G, Hulet C. Reduced wear in vitamin E-infused highly cross-linked polyethylene cups: 5-year results of a randomized controlled trial. Acta Orthop. 2021 Apr;92(2):151-155. doi: 10.1080/17453674.2020.1852785. Epub 2020 Dec 2. PMID 33263447